CLINICAL TRIAL: NCT04616001
Title: Pilot Study of the Use of IVIG in Patients With Severe COVID-19 Infections Requiring Mechanical Ventilation and to Assess Their Biological Responses to IVIG Therapy
Brief Title: IVIG in Patients With Severe COVID-19 Requiring Mechanical Ventilation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sharp HealthCare (Other)
Responsible Party: Principal Investigator, George Sakoulas, MD, Infectious Disease Specialist, Sharp HealthCare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVID-IVIG VENT; 2010902 (Other: Sharp HealthCare Institutional Review Board (SHC IRB))
Record Dates: First submitted 2020-11-02; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Covid19; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Immunoglobulins, Intravenous; Octagam

STUDY DESIGN:
Intervention Model Description: Open label, single group, pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IVIG (Experimental): IVIG 0.5gram/kg IVPB using actual body weight daily x 4 days
  Interventions: Drug: IVIG

INTERVENTIONS:
Drug: IVIG — Patients will receive IVIG daily for four days.
  Other Names: Octagam

SUMMARY:
The purpose of this Pilot Study is to establish a hypothesis of whether or not intravenous immunoglobulin (IVIG) may impact the hospital length of stay, if started within 48 of mechanical ventilation in patients infected with SARS-CoV-2 virus.

DETAILED DESCRIPTION:
This is an investigator initiated, open label, 1 arm study to observe the impact of length of hospitalization by starting IVIG administration within 48 hours of mechanical ventilation. The exploratory objective is to analyze the blood before, during and after IVIG administration. The blood will be analyzed for the production of inflammatory and non-inflammatory cytokines, biomarkers for endothelial injury and biomarkers for coagulation via Mass Spectrometry.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed COVID-19 positive test result
2. Initiation of the first dose of IVIG within 72 hours of mechanical ventilation.
3. Age >18 years old.
4. Consenting next of kin having access to an electronic device that is able to access DocuSign® online and email for consenting.
5. Subjects or their proxy must have the ability to understand the requirements of the study, provide informed consent, and provide authorization of use and disclosure of personal health information.

Exclusion Criteria:

1. Superimposed bacterial pneumonia or bacteremia
2. Severe allergy to any IVIG product formulation
3. Hypersensitivity to corn
4. Uncontrolled hypertension (SBP>180 mm Hg or DBP>120mmHg)
5. Active participant in another research treatment study
6. Advanced dementia
7. Severe renal disease (CrCl< 20 mL/min)
8. Active cancer malignancy
9. Active treatment with cancer chemotherapy or immunotherapy
10. Congestive heart failure clinically or by history (EF< 25%)
11. Prior receipt during admission of any other investigational agent (eg. convalescent plasma, tocilizumab)
12. Venous or arterial thrombosis < 90 days prior
13. Are receiving cytotoxic or biologic treatments such as TNF inhibitors, anti-interleukin-1 (IL-1), anti-IL-6 (tocilizumab or sarilumab), T-cell or B-cell targeted therapies (rituximab), interferon, or Janus kinase (JAK) inhibitors for any indication at study entry. Note: A washout period 4 weeks (or 5 half-lives, whichever is longer) is required prior to screening, with the following exceptions:

    * B-cell targeted therapies: a washout period of 24 weeks or 5 half-lives (whichever is longer)
    * TNF inhibitors: a washout period of 2 weeks or 5 half-lives (whichever is longer), and
    * JAK inhibitor: a washout period of 1 week or 5 half-lives (whichever is longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | Up to 60 days
  Assess hospital length of stay after mechanical ventilation

SECONDARY OUTCOMES:
Human metabolome and proteome | Up to 60 days
  Analyze the blood to assess the human metabolome and proteome in patients with COVID-19 receiving IVIG including production of inflammatory and anti-inflammatory cytokines, markers of endothelial injury, and coagulation using Mass Spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: George Sakoulas, MD, Principal Investigator — Sharp HealthCare
Locations (1):
- Sharp Memorial Hospital, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No